CLINICAL TRIAL: NCT01203709
Title: Low-dose Combination of Mycophenolate Mofetil and Tacrolimus for Refractory Lupus Nephritis: a 12-month Prospective Study
Brief Title: Low-dose Combination of Mycophenolate Mofetil (MMF) and Tacrolimus (Tac) for Refractory Lupus Nephritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Consultant, Tuen Mun Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTWC/CREC/837/10
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Lupus Nephritis
Keywords: lupus; nephritis; glomerulonephritis; nephropathy; refractory
MeSH Terms: conditions — Lupus Nephritis; Nephritis; Glomerulonephritis; Kidney Diseases | interventions — Triamcinolone; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination treatment (Experimental): treatment arm
  Interventions: Drug: low dose combination of MMF and Tac

INTERVENTIONS:
Drug: low dose combination of MMF and Tac — mycophenolate mofetil 500mg BID + tacrolimus 2mg BID
  Other Names: Cellcept and Prograf

SUMMARY:
A trial of combination of two drugs for the treatment of refractory lupus nephritis.

DETAILED DESCRIPTION:
Low-dose combination of mycophenolate mofetil and tacrolimus for refractory lupus nephritis: a 12-month prospective study

ELIGIBILITY:
Inclusion Criteria:

1. Active nephritis documented by renal biopsy within 24 months of entry;
2. Failure to respond to 2 or more immunosuppressive regimens which consisted of high-dose prednisolone combined with other non-corticosteroid immunosuppressive agents together with ACE inhibitors plus or minus angiotensin receptor blockers (ARB) for at least 4 months for each regimen at the maximally tolerated drug dosages;
3. Serum creatinine (Scr) less than 200umol/L.

Exclusion Criteria:

1. Previous intolerance to either MMF/Tac;
2. Scr >200umol/L;
3. Informed consent unavailable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Clinical remission rate | 12 months

SECONDARY OUTCOMES:
Adverse events | 12 months
  adverse events experienced by patients as a measure of tolerability

CONTACTS AND LOCATIONS:
Overall Officials: CC Mok, MD, FRCP, Principal Investigator — Tuen Mun Hospital, Hong Kong China
Locations (1):
- Tuen Mun Hospital, Hong Kong, China